CLINICAL TRIAL: NCT05924386
Title: Marginal Bone Changes in Fixed All-on-Four Mandibular Prosthesis Using OT Bridge Attachment System Versus Conventionally Screw Retained Multiunit Abutments: A Randomized Clinical Trial
Brief Title: Marginal Bone Changes in Fixed All-on-Four Mandibular Prosthesis Using OT Bridge Attachment System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, Nesma osama, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4223
Record Dates: First submitted 2023-06-06; First posted 2023-06-29 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Jaw
Keywords: OTbridge attachment; ALL ON 4; fixed supported implant prosthesis; conventional screw retained fixed prosthesis
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: edentulous patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- All-on-four fixed mandibular prosthesis using conventionally screw retained multiunit abutments. (Active Comparator): Edentulous patients receiving All-on-four fixed mandibular prosthesis using conventionally screw retained multiunit abutments.
  Interventions: Procedure: patients reciveing all on 4 fixed mandibular prosthesis usimg conventionally screw retained multiunit abutments
- All-on-four fixed mandibular prosthesis using OT bridge attachment system (Experimental): Edentulous patients receiving All-on-four fixed mandibular prosthesis using OT bridge attachment system
  Interventions: Procedure: all on 4 fixed mandibular prosthesis using OTbridge attachment system

INTERVENTIONS:
Procedure: patients reciveing all on 4 fixed mandibular prosthesis usimg conventionally screw retained multiunit abutments — Multiunit abutments is considered a gold standard screw retained abutments. Multi-unit abutments are used to correct for varying heights among the implants, to establish a level restorative platform for the prosthesis, as well as to situate the implant connection even with or just below the gingival surface. Also they are used to correct the angulation of implants, helping to keep the screw access holes away from the facial surfaces of the restoration, and facilitate the path of insertion of prosthesis.
  Arms: All-on-four fixed mandibular prosthesis using conventionally screw retained multiunit abutments.
Procedure: all on 4 fixed mandibular prosthesis using OTbridge attachment system — The OT bridge attachment system introduced by (Rhein 83) is a global, well-established system used in the removable prosthetic protocols, the presence of seeger acetal ring placed between the sub-equatorial area of the OT Equator and the cylindrical "Extragrade" abutment compensates the space between the extragrade abutment and the OT equator attachment correcting the minor misalignments that produced during the prosthetic procedure and resulting in more passive fit.
  Arms: All-on-four fixed mandibular prosthesis using OT bridge attachment system

SUMMARY:
Group I (control) Edentulous mandible receiving all on four fixed mandibular prosthesis using conventionally screw retained multiunit abutments.

Group II (intervention) Edentulous mandible receiving all on four fixed prostheses using OT bridge attachments system.

For both groups, the implant sites will be prepared aided by the surgical template. 4 implants with length 11-13 mm will be placed, two anterior implants will be aligned in an axial orientation and two posterior implants will be distally aligned according to the all-on-four concept in the inter foraminal area. Implants will be ideally placed at bone level.

For both groups:

After implant placement and surgical guide removal, healing abutments ( will be connected during healing periods (eight to twelve weeks).

Group I ( control) After eight to twelve weeks from implant placement, multiunit abutments with appropriate heights and angulations will be connected to the implants.

Group II ( intervention) After eight to twelve weeks from implant placement, narrow- and low-profile OT Equator abutment will be screwed onto the implants according to the manufacturer.

marginal bone changes and prosthetic complications are the outcomes Radiographic follow up will be performed for marginal bone changes Serial of standardized digital periapical radiographs using will be taken at the time fixed prosthesis insertion (baseline), 3,6,9,12 months.

Type and incidence of prosthetic complications for the prothesis for each group will be evaluated in 3, 6,9 and 12 months, these complications included: loosening or fracture of the prosthetic screw, prosthesis mobility and fracture of the prosthesis.

DETAILED DESCRIPTION:
Interventions will be conducted by principal investigator (N.O)

General operative procedures:

Eligible patients will be selected from outpatient clinic in prosthodontic department clinic. Patients Will be informed of the research work and informed consent will be obtained from each patient. Only motivated patients who show cooperation and has all the included criteria will be into the study.

Group I (Control):

Edentulous mandible receiving all on four fixed mandibular prosthesis using conventionally screw retained multiunit abutments.

Group II (intervention):

Edentulous mandible receiving all on four fixed prostheses using OT bridge attachments system.

For both groups, a lower removable complete denture will be constructed for each eligible patient. The lower denture will be duplicated into clear acrylic resin which will be modified with radiopaque markers at the proposed implant sites. This clear stent will function as the scan appliance for CBCT scan for detecting the bone high and width, and for implant planning.

Surgical phase:

All patients in both groups will receive prophylactic antibiotic therapy: 2 g of amoxicillin (or clindamycin 600 mg if allergic to penicillin) 1 h before the intervention and rinse with chlorhexidine mouthwash 0.2% for one minute prior to the intervention. The implants will be placed with a fully surgical guided template, under local anesthesia (artcaine with adrenaline 1:100,000), and according to the manufacturer's instructions.

For both groups, the implant sites will be prepared aided by the surgical template. 4 implants (Neobiotech Co.,Ltd, Korea) with length 11-13mm will be placed, two anterior implants will be aligned in an axial orientation and two posterior implants will be distally aligned according to the all-on-four concept in the inter foraminal area. The standard sequence of the osteotomy site preparation will be followed to accommodate the selected implant size. Implants will be ideally placed at bone level.

Page 12 of 22 Group I: After implant placement and surgical guide removal, screwed healing abutments (Neobiotech Co.,Ltd, Korea) will be connected during healing periods (eight to twelve weeks).

Group II: After implant placement and surgical guide removal, screwed healing abutments of (Rhien'83) will be connected during the healing period (eight to twelve weeks).

After the surgical procedures end, all the patients will receive drugs prescription, oral and written recommendations about the correct oral hygiene maintenance and diet.

Prosthetic phase:

Group I:

After eight to twelve weeks from implant placement, multiunit abutments (Neobiotech Co.,Ltd, Korea) with appropriate heights and angulations will be connected to the implants. Impressions will be taken using open tray impression technique for construction of framework superstructure, a posterior cantilever extended to the first molar tooth. The passivity of the metallic framework will be validated intraorally by means of using the single screw test. The non-passive fit will be corrected by sectioning and soldering. The acrylic veneering of the metal superstructure will be made.

Group II:

After eight to twelve weeks from implant placement, narrow- and low-profile OT Equator abutments (Rhein'83, Bologna, Italy) will be screwed onto the implants according to the manufacturer. The trans-mucosal height of the abutments will be chosen based on the soft tissue thickness and implant depth. Impressions will be taken using open tray impression technique for construction of framework superstructure a posterior cantilever extended to the first molar tooth. the cast framework superstructure splinting all implants will be constructed after placing the acetal rings (Seeger system, Rhein'83) between the subequatorial area of the OT Equators (Rhein'83) and the cylindrical "extra grade" framework connections. Then the prosthesis will be screwed twice at 20 N For both groups, occlusion will be checked using articulating paper for any occlusal interferences, and patients will be enrolled in a strictly follow-up protocol including occlusal adjustment and hygiene maintenance every 3 months.

Outcomes:

Primary outcome Marginal bone loss will be measured by using periapical X-ray with parallel technique (Digora system), unit of measurment is Millimeter.

Prosthetic complications as:

1. Loosening of prosthetic screw
2. Fracture of prosthetic screw
3. Prosthesis fracture These outcomes are Binary and will be measure if incidence of complication happened or not by using (Yes/No).

Primary outcome:Radiographic follow up will be performed for marginal bone changes. Serial of standardized digital periapical radiographs using; long cone paralleling technique, XCP periapical film holder and an individually constructed radiographic acrylic template will be taken at the time fixed prosthesis insertion (baseline), 3,6,9,12 months.

The software of the Digora system will be used for evaluation of the marginal bone changes. Lines parallel to the long axis of the mesial and distal surface of each abutment will be made. The distance in mm from the crest of alveolar bone to the apex of the tooth will be measured and the marginal bone changes in the subsequent measurements will be calculated.

Secondary outcome:

Type and incidence of prosthetic complications for the prothesis for each group will be evaluated in 3, 6,9 and 12 months, these complications included: loosening or fracture of the prosthetic screw, prosthesis mobility and fracture of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

Patients with completely edentulous patients

* Aged 40 years or older.
* Sufficient inter -arch space not less than 13 mm.
* Good oral hygiene
* Minimum bone height 10 mm and minimum bone diameter should be 6 mm

Exclusion Criteria:

* General contraindications for oral surgery
* Heavy smokers (greater than 20 cigarettes a
* Local acute or chronic infections
* Substance abuse (drugs or alcohol)
* Patients with neuromuscular or psychiatric disorders.
* Treatment with intravenous bisphosphonates
* Irradiation of the neck or head area in the past 5 years
* Diabetic patients (HbA1c>7.5%)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss | 1 year follow up
  Radiographic follow up will be performed for marginal bone changes. Serial of standardized digital periapical radiographs using; long cone paralleling technique, XCP periapical film holder and an individually constructed radiographic acrylic template will be taken at the time fixed prosthesis insertion (baseline), 3,6,9,12 months.
  The software of the Digora system will be used for evaluation of the marginal bone changes. Lines parallel to the long axis of the mesial and distal surface of each abutment will be made. The distance in mm from the crest of alveolar bone to the apex of the tooth will be measured and the marginal bone changes in the subsequent measurements will be calculated.

SECONDARY OUTCOMES:
prosthetic complications | 1 year follow up
  Type and incidence of prosthetic complications for the prothesis for each group will be evaluated in 3, 6,9 and 12 months, these complications included: loosening or fracture of the prosthetic screw, prosthesis mobility and fracture of the prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: nesma O elmosallamy, Principal Investigator — CAIRO UNIVERISTY
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No